CLINICAL TRIAL: NCT03820583
Title: Whipple Procedure: A 5-year Clinical Experience in Tertiary Care Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Principle investigator, Services Hospital, Lahore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s11
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Whipple Procedure
Keywords: Whipple procedure, pancreatic carcinoma, biliary stenting,
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Intervention Model Description: Patients undergoing Whipple procedure due to pancreatic tumor were included in the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Whipple Procedure — Patients underwent Whipple procedure for pancreatic tumors. The procedure commenced with rooftop incision. then layers of abdomen dissected to reach the peritoneum. Then Duodenum dissected out along with pancreas and common bile duct. After rescetion of these structures the anatomy of the tract restored with three anastomosis namely pancreaticojejunostomy, gastrojejunostomy and choledochojejunostomy/hepaticojejunostomy.

SUMMARY:
The study was conducted in tertiary care hospital of Lahore. Patient undergoing Whipple procedure were studied by compiling demographic details of the patients, common presenting symptoms, various indications for Whipple's procedure, the cofactors which affect the procedures outcome and morbidity and mortality of the patients.

DETAILED DESCRIPTION:
This study was performed by collecting data through predesigned questionnaire about patients undergoing Whipple's procedure from operation theatres and medical record section. Those patients, whose tumor was unresectable and undergone palliative surgical procedures were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* patients of both sexes with age ranging from 20 years to 70 years
* patients with pancreatic tumors
* patients with adequate cardiorespiratory reserves to be fit for prolong general anesthesia

Exclusion Criteria:

* unresectable tumors
* unfit for surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients developing pancreatic fistula | 4 weeks
  Percentage of patients developing pancreatic fistula (pancreatic juice collected in drain rich in amylase) after Whipple procedure Enteric leak postoperative complications like pancreatic fistula, anastomotic leakage, hemorrhage, wound infection,mortality
Percentage of patients developing hemorrhage | 2 weeks
  Percentage of patients developing hemorrhage after Whipple procedure
Percentage of patients developing wound infection | 4 weeks
  Percentage of patients developing wound infection after Whipple procedure
Mortality rate | 6 weeks
  Mortality of patients undergoing Whipple surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mahmmood Ayyaz, mbbs, fcps, Study Director — Services Hospital, Lahore
Locations (1):
- Services hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided